CLINICAL TRIAL: NCT01753193
Title: A Phase 2, Open-label Extension Study to Evaluate Long-term Safety of MEDI-546 in Adults With Systemic Lupus Erythematosus
Brief Title: An Open-label Study to Evaluate the Long-term Safety of MEDI-546, for the Treatment of SLE, in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD-IA-MEDI-546-1145; 2012-004619-30 (EudraCT Number)
Record Dates: First submitted 2012-12-17; First posted 2012-12-20 (Estimated); Results first posted 2019-07-31 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — anifrolumab

STUDY DESIGN:
Intervention Model Description: This is an Open Label Extension study.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Anifrolumab (Experimental): Participants will receive IV infusion of anifrolumab 1000 milligrams (mg) every 4 weeks (Q4W) from Day 1 (Week 0) until 12-Feb-2015 (approval of protocol amendment 4); and thereafter will receive 300 mg Q4W for up to 3 years or until the sponsor discontinued development of anifrolumab, whichever came first.
  Interventions: Biological: Anifrolumab

INTERVENTIONS:
Biological: Anifrolumab — Intravenous infusion of anifrolumab will be administered as 1000 mg Q4W from Day 1 (Week 0) until 12-Feb-2015 (approval of protocol amendment 4); and thereafter 300 mg Q4W up to 3 years or until the sponsor discontinued development of anifrolumab, whichever came first.
  Other Names: MEDI-546

SUMMARY:
The purpose of this study is to evaluate the long-term safety of anifrolumab (MEDI-546) in adults with moderate to severe active systemic lupus erythematosus (SLE).

DETAILED DESCRIPTION:
This is an open-label extension study to evaluate long-term safety and tolerability of intravenous (IV) anifrolumab in adult participants with moderately-to-severely active SLE. Participants must have completed the qualifying Phase 2 study and meet this study criteria in order to be eligible.

ELIGIBILITY:
Inclusion Criteria:

* Must be willing to use 2 methods of effective contraception
* Must have venous access
* Must be willing to forego participation in other clinical trials for SLE.

Exclusion Criteria:

* Any concurrent condition that in the opinion of the investigator would interfere with the evaluation of the investigational product
* Major surgery within 8 weeks before signing informed consent form (ICF)
* Elective major surgery planned during the study period
* Concomitant Medications within the last 12 weeks: Azathioprine > 200 mg/day, Mycophenolate mofetil/mycophenolic acid > 2.0 g/day, oral, subcutaneous, or intramuscular methotrexate > 25 mg/week
* A live or attenuated vaccine within 4 weeks of signing the ICF
* Bacillus of Calmette and Guérin (BCG) vaccine within 1 year of ICF

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2013-03-28 (Actual); Primary Completion 2018-07-18 (Actual); Study Completion 2018-07-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (55):
- United States (22):
  - Research Site, Birmingham, Alabama
  - Research Site, La Palma, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Palm Desert, California
  - Research Site, Upland, California
  - Research Site, Ocala, Florida
  - Research Site, Orlando, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Stockbridge, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Las Cruces, New Mexico
  - Research Site, New York, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Tulsa, Oklahoma
  - Research Site, Memphis, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Spokane, Washington
- Brazil (2):
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
- Bulgaria (2):
  - Research Site, Plovdiv
  - Research Site, Sofia
- Colombia (5):
  - Research Site, Barranquilla
  - Research Site, Bogotá
  - Research Site, Bucaramanga
  - Research Site, Chía
  - Research Site, Medellín
- Czechia (2):
  - Research Site, Brno
  - Research Site, Prague
- Research Site, Debrecen, Hungary
- Mexico (4):
  - Research Site, Guadalajara
  - Research Site, León
  - Research Site, México
  - Research Site, Toluca
- Peru (2):
  - Research Site, Arequipa
  - Research Site, Lima
- Poland (4):
  - Research Site, Bialystok
  - Research Site, Krakow
  - Research Site, Nadarzyn
  - Research Site, Poznan
- Research Site, Iași, Romania
- South Korea (3):
  - Research Site, Gwangju
  - Research Site, Seodaemun-gu
  - Research Site, Suwon
- Taiwan (2):
  - Research Site, Chiayi City
  - Research Site, Zhongzheng District
- Ukraine (5):
  - Research Site, Donetsk
  - Research Site, Kyiv
  - Research Site, Ternopil
  - Research Site, Vinnitsya
  - Research Site, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
AstraZeneca's policy is to share data with researchers if the request is in scope of our policy. Additional information can be found on astrazenecaclinicaltrials.com.

REFERENCES:
- [Derived] Chatham WW, Furie R, Saxena A, Brohawn P, Schwetje E, Abreu G, Tummala R. Long-Term Safety and Efficacy of Anifrolumab in Adults With Systemic Lupus Erythematosus: Results of a Phase II Open-Label Extension Study. Arthritis Rheumatol. 2021 May;73(5):816-825. doi: 10.1002/art.41598. Epub 2021 Mar 24. PMID 33225631

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 28 Mar 2013 to 18 Jul 2018.
Pre-assignment Details: A total of 218 participants were enrolled in this open-label extension (OLE) study.
Groups:
- Anifrolumab: Participants received intravenous (IV) infusion of anifrolumab (MEDI-546) 1000 milligrams (mg) every 4 weeks (Q4W) from Day 1 (Week 0) until 12-Feb-2015 (approval of protocol amendment 4); and thereafter received 300 mg Q4W for up to 3 years or until the sponsor discontinued development of anifrolumab, whichever came first.
Period: Overall Study
Arm/Group | Anifrolumab
Started | 218
Completed | 172
Not Completed | 46
Not completed — Withdrawal by Subject | 23
Not completed — Lost to Follow-up | 6
Not completed — Death | 1
Not completed — Other | 16

BASELINE CHARACTERISTICS:
Population: As-treated population included all participants who received any dose of study drug in the OLE study.
Arm/Group | Anifrolumab
Number analyzed (Participants) | 218
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.8 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 203
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 104
  Not Hispanic or Latino | 114
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 29
  White | 87
  More than one race | 2
  Unknown or Not Reported | 85

OUTCOME MEASURES:

1. Primary Outcome: Number of Particpants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event is any AE that resulted in death, life threatening, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, is a congenital anomaly/birth defect in offspring of a study participant, is an important medical event that may jeopardize the participant or may require medical intervention. TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: From first dose of study drug (Day 1) through 168 weeks
Population: As-treated population included all participants who received any dose of study drug in the OLE study.
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab
Number analyzed (Participants) | 218
Participants
  TEAEs | 170
  TESAEs | 50

2. Primary Outcome: Number of Participants With Adverse Events Resulting in Discontinuation (DAEs) of Anifrolumab
Description: Number of participants with DAEs are reported.
Time Frame: From first dose of study drug (Day 1) through 168 weeks
Population: As-treated population included all participants who received any dose of study drug in the OLE study.
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab
Number analyzed (Participants) | 218
Participants | 17

3. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibodies (ADA) Titer to Anifrolumab
Description: The number of participants with positive serum antibodies to anifrolumab at anytime (including baseline) are reported.
Time Frame: Baseline (Pre-dose on Day 1) up to Week 168
Population: As-treated population included all participants who received any dose of study drug in the OLE study. Participants with reportable ADA titer results were analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab
Number analyzed (Participants) | 216
Participants | 5

4. Secondary Outcome: Anti-Drug Antibodies (ADA) Titer to Anifrolumab
Description: Median ADA titer in participants with ADA-positive assessments and reportable ADA titer results are reported.
Time Frame: Baseline (Pre-dose on Day 1) up to Week 168
Population: As-treated population included all participants who received any dose of study drug in the OLE study. Only participants who had ADA-positive assessments with reportable ADA titer results were analyzed for this outcome measure.
Measure: Median (Full Range); unit: Antibody titers
Arm/Group | Anifrolumab
Number analyzed (Participants) | 5
Antibody titers | 120 [30 to 120]

5. Secondary Outcome: Number of ADA-positive Participants With Decreased Serum Concentration of Anifrolumab
Description: Number of participants with decreased serum concentration of anifrolumab due to ADA-positive results are reported.
Time Frame: Baseline (Pre-dose on Day 1) up to Week 168
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab
Number analyzed (Participants) | 5
Participants | 1

6. Secondary Outcome: Number of ADA-positive Participants With Decreased Pharmacodynamics Response of Anifrolumab
Description: Number of participants with decreased pharmacodynamic response of anifrolumab due to ADA-positive results are reported.
Time Frame: Baseline (Pre-dose on Day 1) up to Week 168
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab
Number analyzed (Participants) | 5
Participants | 1

7. Secondary Outcome: Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) Global Score for ADA Positive Participants
Description: The SLEDAI-2K is an activity index that measures disease activity and records feature of active lupus as present or not present. SLEDAI-2K uses a weighted checklist to assign a numerical score based on the presence or absence of 24 symptoms. Each symptom present is assigned between 1 and 8 points based on its usual clinical importance, yielding a total score that ranges from 0 points (no symptoms) to 105 points (presence of all defined symptoms).
Time Frame: Baseline (Pre-dose on Day 1); and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 160, and 168
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on Score
Arm/Group | Anifrolumab
Number analyzed (Participants) | 5
Units on Score
  Baseline | 7.8 (7.6)
  Week 12: number analyzed (Participants) | 4
  Week 12 | 5 (2.0)
  Week 24: number analyzed (Participants) | 4
  Week 24 | 1.5 (1.9)
  Week 36: number analyzed (Participants) | 4
  Week 36 | 2.0 (2.3)
  Week 48 | 1.8 (2.0)
  Week 60: number analyzed (Participants) | 4
  Week 60 | 2.0 (1.6)
  Week 72: number analyzed (Participants) | 2
  Week 72 | 4.0 (5.7)
  Week 84: number analyzed (Participants) | 2
  Week 84 | 3.0 (1.4)
  Week 96: number analyzed (Participants) | 2
  Week 96 | 3.0 (1.4)
  Week 108: number analyzed (Participants) | 2
  Week 108 | 4.0 (0.0)
  Week 120: number analyzed (Participants) | 2
  Week 120 | 5.0 (1.4)
  Week 132: number analyzed (Participants) | 2
  Week 132 | 4.0 (0.0)
  Week 144: number analyzed (Participants) | 2
  Week 144 | 7.0 (7.1)
  Week 156: number analyzed (Participants) | 2
  Week 156 | 6.0 (2.8)
  Week 160: number analyzed (Participants) | 2
  Week 160 | 2.0 (2.8)
  Week 168: number analyzed (Participants) | 2
  Week 168 | 2.0 (2.8)

8. Secondary Outcome: Number of ADA-positive Participants With TEAEs and TESAEs
Description: The number of ADA-positive participants with TEAEs and TESAEs are reported.
Time Frame: Baseline (Pre-dose on Day 1) up to Week 168
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab
Number analyzed (Participants) | 5
Participants
  TEAEs | 5
  TESAEs | 1

9. Primary Outcome: Number of Participants With Adverse Events of Special Interest (AESIs)
Description: An AESI is scientific and medical concern specific to understanding of the study drug. An AESI may be serious or non-serious. Number of participants with AESIs are reported.
Time Frame: From first dose of study drug (Day 1) through 168 weeks
Population: As-treated population included all participants who received any dose of study drug in the OLE study.
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab
Number analyzed (Participants) | 218
Participants
  Herpes zoster | 11
  Drug hypersensitivity | 1
  Hypersensitivity | 2
  Infusion related reaction | 4
  Nausea | 1
  Hodgkin's disease | 1
  Latent tuberculosis | 5
  Hypersensitivity vasculitis | 1
  Vasculitis | 1

ADVERSE EVENTS:
Time Frame: From first dose of study drug (Day 1) through 168 weeks
Arm/Group | Anifrolumab
All-Cause Mortality (participants affected / at risk) | 1/218
Serious Adverse Events (participants affected / at risk) | 50/218
Other Adverse Events (participants affected / at risk) | 164/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anifrolumab (N=218)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (2)
Cardiac failure (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Hypothalamic pituitary adrenal axis suppression (Endocrine disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Cyst (General disorders) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1)
Chikungunya virus infection (Infections and infestations) | 2 (2)
Dengue fever (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2)
Herpes zoster (Infections and infestations) | 1 (1)
Latent tuberculosis (Infections and infestations) | 1 (1)
Mastoiditis (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 4 (5)
Pneumonia bacterial (Infections and infestations) | 1 (1)
Post procedural infection (Infections and infestations) | 2 (2)
Pyelonephritis (Infections and infestations) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 (3)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 5 (5)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (2)
Dizziness (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Idiopathic intracranial hypertension (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (2)
Syncope (Nervous system disorders) | 1 (1)
High risk pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 2 (2)
Renal impairment (Renal and urinary disorders) | 1 (1)
Cervical polyp (Reproductive system and breast disorders) | 1 (1)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 2 (2)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anifrolumab (N=218)
Anaemia (Blood and lymphatic system disorders) | 6 (6)
Hypercoagulation (Blood and lymphatic system disorders) | 1 (1)
Hyperleukocytosis (Blood and lymphatic system disorders) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Leukaemoid reaction (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 2 (6)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Neutrophilia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (2)
Angina pectoris (Cardiac disorders) | 2 (2)
Bifascicular block (Cardiac disorders) | 2 (2)
Bundle branch block right (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Left atrial dilatation (Cardiac disorders) | 1 (1)
Myocardial fibrosis (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 2 (2)
Ventricular extrasystoles (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 2 (2)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 1 (1)
Hyperparathyroidism primary (Endocrine disorders) | 1 (1)
Thyroid mass (Endocrine disorders) | 1 (1)
Blepharitis (Eye disorders) | 1 (1)
Blepharochalasis (Eye disorders) | 2 (2)
Cataract (Eye disorders) | 4 (4)
Chalazion (Eye disorders) | 1 (1)
Eyelid oedema (Eye disorders) | 1 (1)
Macular degeneration (Eye disorders) | 1 (1)
Myopia (Eye disorders) | 1 (1)
Scleritis (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Visual acuity reduced (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (3)
Abdominal pain upper (Gastrointestinal disorders) | 5 (6)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 5 (5)
Dental caries (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 11 (12)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1)
Gastric mucosa erythema (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 2 (2)
Gastritis (Gastrointestinal disorders) | 7 (7)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Internal hernia (Gastrointestinal disorders) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (8)
Noninfective gingivitis (Gastrointestinal disorders) | 1 (1)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Acquired gene mutation (General disorders) | 1 (1)
Asthenia (General disorders) | 4 (4)
Cyst (General disorders) | 1 (1)
Influenza like illness (General disorders) | 6 (10)
Oedema peripheral (General disorders) | 4 (4)
Pyrexia (General disorders) | 5 (5)
Tenderness (General disorders) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 3 (3)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 2 (3)
Hypersensitivity (Immune system disorders) | 2 (2)
Seasonal allergy (Immune system disorders) | 2 (2)
Acarodermatitis (Infections and infestations) | 1 (1)
Acute sinusitis (Infections and infestations) | 2 (2)
Appendicitis (Infections and infestations) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 2 (2)
Body tinea (Infections and infestations) | 1 (1)
Bone abscess (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 28 (33)
Bronchitis bacterial (Infections and infestations) | 1 (1)
Bronchitis viral (Infections and infestations) | 1 (1)
Candida infection (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 3 (8)
Cervicitis (Infections and infestations) | 2 (2)
Conjunctivitis (Infections and infestations) | 3 (3)
Cystitis (Infections and infestations) | 3 (3)
Dermatophytosis of nail (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 2 (2)
Furuncle (Infections and infestations) | 3 (4)
Gastroenteritis (Infections and infestations) | 5 (6)
Gastroenteritis viral (Infections and infestations) | 4 (4)
Gastrointestinal viral infection (Infections and infestations) | 1 (1)
Genital candidiasis (Infections and infestations) | 1 (1)
Genital herpes simplex (Infections and infestations) | 1 (1)
Herpes simplex (Infections and infestations) | 2 (2)
Herpes zoster (Infections and infestations) | 10 (10)
Infected bite (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 9 (10)
Latent tuberculosis (Infections and infestations) | 5 (5)
Lymphangitis (Infections and infestations) | 1 (1)
Nail infection (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 32 (40)
Onychomycosis (Infections and infestations) | 1 (1)
Oral candidiasis (Infections and infestations) | 2 (3)
Oral herpes (Infections and infestations) | 6 (7)
Oropharyngeal candidiasis (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 4 (4)
Papilloma viral infection (Infections and infestations) | 1 (1)
Paronychia (Infections and infestations) | 2 (2)
Parotitis (Infections and infestations) | 1 (1)
Pelvic inflammatory disease (Infections and infestations) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 10 (11)
Pharyngitis streptococcal (Infections and infestations) | 3 (3)
Pharyngotonsillitis (Infections and infestations) | 2 (2)
Pleurisy viral (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 4 (6)
Pneumonia bacterial (Infections and infestations) | 1 (1)
Pulpitis dental (Infections and infestations) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 8 (12)
Skin candida (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Streptococcal infection (Infections and infestations) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 2 (3)
Tinea manuum (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 3 (3)
Tracheobronchitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 20 (29)
Urinary tract infection (Infections and infestations) | 13 (17)
Urinary tract infection fungal (Infections and infestations) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 5 (5)
Viral upper respiratory tract infection (Infections and infestations) | 5 (6)
Vulval abscess (Infections and infestations) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 2 (2)
Vulvovaginal mycotic infection (Infections and infestations) | 3 (3)
Vulvovaginitis (Infections and infestations) | 1 (1)
Zika virus infection (Infections and infestations) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 5 (5)
Epicondylitis (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 4 (9)
Injection related reaction (Injury, poisoning and procedural complications) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 4 (5)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Scar (Injury, poisoning and procedural complications) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood immunoglobulin a decreased (Investigations) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1)
Electrocardiogram qt shortened (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)
Lipids abnormal (Investigations) | 1 (1)
Liver function test increased (Investigations) | 2 (2)
Mycobacterium tuberculosis complex test positive (Investigations) | 1 (1)
Neutrophil count increased (Investigations) | 2 (4)
Nuclear magnetic resonance imaging brain abnormal (Investigations) | 1 (1)
Transaminases increased (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Weight increased (Investigations) | 1 (1)
Acquired mixed hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (6)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Vitamin d deficiency (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (8)
Bursitis (Musculoskeletal and connective tissue disorders) | 2 (2)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteochondritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 (4)
Osteopenia (Musculoskeletal and connective tissue disorders) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 3 (4)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (3)
Haemangioma of bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Vulvovaginal warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Cerebrovascular disorder (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 5 (6)
Encephalopathy (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 14 (21)
Hypersomnia (Nervous system disorders) | 1 (1)
Intercostal neuralgia (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Lumbosacral radiculopathy (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 4 (6)
Paraesthesia (Nervous system disorders) | 1 (1)
Pineal gland cyst (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 4 (4)
Visual field defect (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 4 (4)
Libido decreased (Psychiatric disorders) | 2 (2)
Dysuria (Renal and urinary disorders) | 1 (1)
Hypertonic bladder (Renal and urinary disorders) | 1 (1)
Nephritis (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Breast discharge (Reproductive system and breast disorders) | 1 (2)
Breast tenderness (Reproductive system and breast disorders) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1)
Cervical polyp (Reproductive system and breast disorders) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1)
Dyspareunia (Reproductive system and breast disorders) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1)
Endometrial thickening (Reproductive system and breast disorders) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Menometrorrhagia (Reproductive system and breast disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Menstruation delayed (Reproductive system and breast disorders) | 1 (1)
Menstruation irregular (Reproductive system and breast disorders) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Polymenorrhoea (Reproductive system and breast disorders) | 1 (1)
Uterine cervical erosion (Reproductive system and breast disorders) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1)
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 (1)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1)
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 1 (1)
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 1 (1)
Idiopathic urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 1 (1)
Mechanical urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Panniculitis (Skin and subcutaneous tissue disorders) | 3 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (3)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (4)
Hypertension (Vascular disorders) | 3 (3)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (2)
Peripheral coldness (Vascular disorders) | 1 (2)
Peripheral venous disease (Vascular disorders) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1)
Raynaud's phenomenon (Vascular disorders) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises on going studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2015-02-12): https://cdn.clinicaltrials.gov/large-docs/93/NCT01753193/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/93/NCT01753193/SAP_001.pdf